CLINICAL TRIAL: NCT04960696
Title: An Evaluation of the Effect on Ocular Surface Symptoms of Online Education During the Pandemic
Brief Title: Effect on Ocular Surface Symptoms of Online Education
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Abdullah Beyoğlu, Assist of Prof, Kahramanmaras Sutcu Imam University
Other Study IDs: desicion:06, dated: 12/04/21
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Eye Diseases; Ocular Surface Disease; Dry Eye
Keywords: Pandemic; online education; ocular health; tear break up time; schirmer
MeSH Terms: conditions — Eye Diseases; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- primary school/78 subjects: Determining the negative effects of distance education on eye symptoms during the pandemic period.
  Interventions: Diagnostic Test: OSDI; Diagnostic Test: tear break up time; Diagnostic Test: schirmer
- middle school/78 subjects: Determining the negative effects of distance education on eye symptoms during the pandemic period.
  Interventions: Diagnostic Test: OSDI; Diagnostic Test: tear break up time; Diagnostic Test: schirmer
- high school/78 subjects: Determining the negative effects of distance education on eye symptoms during the pandemic period.
  Interventions: Diagnostic Test: OSDI; Diagnostic Test: tear break up time; Diagnostic Test: schirmer
- university/81 subjects: Determining the negative effects of distance education on eye symptoms during the pandemic period.
  Interventions: Diagnostic Test: OSDI; Diagnostic Test: tear break up time; Diagnostic Test: schirmer

INTERVENTIONS:
Diagnostic Test: OSDI — Change of OSDI in distance education
Diagnostic Test: tear break up time — Change of tear break up time in distance education
Diagnostic Test: schirmer — Change of schirmer in distance education

SUMMARY:
retrospective, observational study.

DETAILED DESCRIPTION:
Aim: The aim of this study was to investigate the effects on ocular surface symptoms of students taking online education, which was a part of the distance learning model during the COVID-19 pandemic, to be able to prevent the formation of irreversible damage with early diagnosis and treatment. With recommendations that can be simply applied, it was aimed to protect ocular health.

Material and Method: The study included 315 students who were undertaking online education and presented at the Ophthalmology Department of a tertiary level university hospital. A record was made of sociodemographic data, Schirmer test results, tear break-up time (TBUT) measurements, and Ocular Surface Disease Index (OSDI) scores. The data were analyzed statistically using SPSS vn. 22.0 software, and a value of p<0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Online education >6 years <30 years student

Exclusion Criteria:

not student not taking online education <6 years >30 years

Ages: 6 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes — 6-30 years
Study Population: Students aged 6-30 who receive online education during the pandemic period
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Dry eye symptom scale: ocular symptom scale index (OSDI) | baseline
  Change of OSDI in distance education
Dry eye symptom scale:Tear break up time (TBUT) | baseline
  Change of tear break up time in distance education
Dry eye scale:Schirmer | baseline
  Change of Schirmer in distance education

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Beyoğlu, Study Chair — Kahramanmaraş Sütçü İmam Üniversitesi Tıp Fakültesi
Locations (1):
- Abdullah Beyoğlu, Kahramanmaraş, In the USA Or Canada, Please Select..., Turkey (Türkiye)